CLINICAL TRIAL: NCT00585910
Title: Efficacy and Safety/Tolerability of OROS MPH (Concerta) Plus Atomoxetine (ATMX) in Children and Adolescents (Age 6-17) With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Study of Atomoxetine and OROS Methylphenidate to Treat Children and Adolescents Ages 6-17 With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Timothy Wilens, MD, MD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-P-002180
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2010-05-10 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; Strattera; Concerta; Atomoxetine; OROS Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Total treatment period is 7 weeks. Atomoxetine treatment will be initiated and maintained for 4 weeks. If the subject is a partial responder to atomoxetine treatment, OROS methylphenidate will then be added to his or her treatment regimen for the final 3 weeks of the study.
  Interventions: Drug: Atomoxetine and OROS Methylphenidate

INTERVENTIONS:
Drug: Atomoxetine and OROS Methylphenidate — Subjects must have at least attempted to tolerate a dose of 1.2 mg/kg of atomoxetine. If tolerated, they must remain on this dose for at least two weeks. OROS methylphenidate will be target dosed and titrated to a maximum dose of 54 mg.
  Other Names: Strattera, Concerta

SUMMARY:
The purpose of this study is to evaluate the safety, effectiveness, and tolerability of atomoxetine and OROS methylphenidate, taken together, in the treatment of ADHD in children and adolescents ages 6-17.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients from 6 to 17 years old.
* Subjects with a DSM-IV diagnosis of ADHD by clinical interview, confirmed by the KSADS-E ADHD module.
* Subject with DSM-IV diagnosis of ADHD without previous treatment.
* Subjects with DSM-IV diagnosis of ADHD with a clinical history of a partial response to ATMX or methylphenidate as monotherapy.
* In phase I, subjects with a CGI-Severity of at least moderate impairment related to their ADHD (CGI >4).
* In phase II, subjects receiving therapeutic doses of ATMX with at least minor improvement in their clinical picture due to the ATMX as determined operationally (CGI-Improvement score indicating at least minor improvement relative to off-drug baseline) will be included.
* In phase II, only subjects receiving ATMX that also have evidence of persistent symptoms of ADHD and impairment related to their ADHD (a CGI-Severity of > minor impairment OR ADHD RS >18; AND GAF score <65) will have Concerta added to their regimen.
* Subjects' parents must provide informed consent and subjects' assent.

Exclusion Criteria:

* Pregnant or nursing females or females not using proper contraception.
* Subjects with a medical condition or treatment that will either jeopardize subject safety or affect the scientific merit of the study.
* Subjects (or their families) who do not appear to be reliable reporters of their condition or who indicate they will not be able to meet the schedule of visits for the duration of the study.
* Subjects with Mental Retardation or Organic Brain Syndromes.
* Subjects who have a lifetime history of a psychotic or bipolar disorder.
* Subjects with recent or current (past 30 days) major depressive disorder or a clinically significant anxiety disorder that would potentially necessitate treatment during the trial. g. Subjects with recent evidence (past 30 days) of suicidality or homicidality will not be enrolled.
* Subjects with a recent history (e.g. three months) of a substance use disorder; or those with a positive urine for substances of abuse will not be enrolled. Subjects will be told that a positive urine for substances of abuse will be disclosed to their parents.
* Subjects taking stimulants or other psychotropics at the time of the evaluation. Subjects will not be discontinued from their current medication regimen (not including ATMX), unless authorized and supervised by their treating physician.
* Treatment of stimulants within one week of the evaluation; tricyclic antidepressants, bupropion, cholinesterase inhibitors, modafinil, clonidine/guanfacine, lithium/anticonvulsants for behavioral control, or serotonin reuptake inhibitors (except fluoxetine) for four weeks prior to entry are prohibited. Treatment with antipsychotics/neuroleptics and fluoxetine for 8 weeks prior to entry are prohibited.
* Subjects using any prescribed or over-the-counter concurrent treatment for ADHD.
* Subjects with a history of a lack of response to either ATMX or methylphenidate.
* Subjects with a history of a serious adverse event to either ATMX or methylphenidate.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wilens, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for this study from Outpatient Psychiatry Clinics, the Clinical Pediatric Psychopharmacology Unit of the MGH, and the MGH's extensive network of partnered institutions. Subjects were recruited from 2004 through 2007.
Pre-assignment Details: Some reasons as to why subjects were excluded from the trial before baselining include: being found ineligible, withdrawing consent, and being lost to follow-up.
Groups:
- Overall Study: Atomoxetine (ATMX) treatment will be initiated and maintained for 4 weeks. If the subject is a partial responder to atomoxetine treatment, OROS methylphenidate (OROS MPH) will then be added to his or her treatment regimen for the final 3 weeks of the study. If the subject is not a partial responder to ATMX, they will end their study participation before entering into the ATMX + OROS MPH phase. Subjects already on ATMX before entering the study can enter directly into the OROS MPH phase of the study. 15 out of 55 completed Phase I only and 10 entered directly into Phase II.
Period: Atomoxetine (ATMX) Alone
Arm/Group | Overall Study
Started | 72 (This is the number of subjects who were exposed to ATMX in Phase I of the study.)
Completed | 55 (Number of subjects who completed Phase I. 15 completed only Phase I. 40 proceeded onto Phase II.)
Not Completed | 17
Period: ATMX + Osmotic-Release Methylphenidate
Arm/Group | Overall Study
Started | 50 (Number of participants to add OROS MPH to their ATMX regimen)
Completed | 41
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 72
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.1 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 50
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Attention Deficit Hyperactivity Disorder Rating Scale (ADHD RS)
Description: The primary outcome was the ADHD rating scale. Change scores for the ADHD Rating Scale (RS), from baseline to endpoint (week 7 or last observation carried forward), were analyzed with paired t-tests and nonparametric Wilcoxon sign-rank tests. The best score is a score of 0 (no ADHD symptoms) and the worst score is the highest score possible (54).
Time Frame: 7 weeks
Population: All analyses were intent to treat, with last observation carried forward.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Overall Study
Number analyzed (Participants) | 50
Units on a Scale | 12.8 (9.7)

2. Secondary Outcome: Clinical Global Impressions - Level of Severity (CGIs) for ADHD and Other Psychiatric Disorders
Description: Secondary analyses allowed us to evaluate the effects of treatment on additional measures of functioning (CGIs for ADHD and other psychiatric disorders). The CGI-Severity scale is as follows: 0 = Not assessed, 1 = normal, not at all ill, 2 = Borderline mentally ill, 3 = Mildly ill, 4 = Moderately Ill, 5 = Markedly Ill, 6 = Severely Ill, 7 = Among the most extremely ill patients.
Time Frame: 7 weeks
Measure: Mean (Full Range); unit: Units on a Scale
Arm/Group | Overall Study
Number analyzed (Participants) | 50
Units on a Scale | 2.7 [2.7 to 3.7]

ADVERSE EVENTS:
Groups:
- ATMX Only: Atomoxetine treatment will be initiated and maintained for 4 weeks. If the subject is not a partial responder to ATMX, they will end their study participation before entering into the ATMX + OROS MPH phase.
- ATMX and OROS MPH: Partial responders to ATMX alone entered into the ATMX and OROS MPH phase. Subjects already on ATMX before entering the study can enter directly into the OROS MPH phase of the study. 15 out of 55 completed Phase I only and 10 entered directly into Phase II.
Arm/Group | ATMX Only | ATMX and OROS MPH
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/50
Other Adverse Events (participants affected / at risk) | 72/72 | 50/50
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ATMX Only (N=72) | ATMX and OROS MPH (N=50)
Loss of Appetite (Gastrointestinal disorders) | 13/67 | 22
Gastro-Intestinal (Gastrointestinal disorders) | 34/67 | 17
Insomnia (General disorders) | 10/67 | 25
Headaches (General disorders) | 19/67 | 11
Irritability (Psychiatric disorders) | 11/67 | 16
Fatigue (General disorders) | 29/67 | 3
Rhinitis (General disorders) | 17/67 | 11

LIMITATIONS AND CAVEATS:
* Open trial so may have been biased;
* Small sample size which may have underestimated findings;
* Used a priori definition of partial response. However, our definition of ATMX partial responders has not been validated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No